CLINICAL TRIAL: NCT05755906
Title: A Randomized, Double-Blind, Parallel Group, Multicenter 12 Week Study to Assess the Efficacy and Safety of Budesonide and Formoterol Fumarate Metered Dose Inhaler Relative to Budesonide Metered Dose Inhaler in Participants With Inadequately Controlled Asthma (LITHOS)
Brief Title: A 12-week Study to Assess the Efficacy and Safety of Budesonide and Formoterol Fumarate Metered Dose Inhaler Relative to Budesonide Metered Dose Inhaler in Participants With Inadequately Controlled Asthma (LITHOS)
Acronym: LITHOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5982C00005; 2021-003334-36 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BFF MDI 160/9.6 μg BID (320/19.2μg/day) (Experimental): Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), BDI (320/19.2μg/day)
  Interventions: Drug: BFF MDI 160/9.6 μg BID (320/19.2μg/day)
- BD MDI 160 μg BID (320 μg/day) (Active Comparator): Budesonide (BD) metered-dose inhaler (MDI), 160 μg BID (320 μg/day)
  Interventions: Drug: BD MDI 160 μg BID (320 μg/day)

INTERVENTIONS:
Drug: BFF MDI 160/9.6 μg BID (320/19.2μg/day) — Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg BID (320/19.2μg/day)
  Other Names: BFF
  Arms: BFF MDI 160/9.6 μg BID (320/19.2μg/day)
Drug: BD MDI 160 μg BID (320 μg/day) — Budesonide (BD) metered-dose inhaler (MDI), 160 μg BID (320 μg/day)
  Other Names: BD
  Arms: BD MDI 160 μg BID (320 μg/day)

SUMMARY:
This is a 12-week study to evaluate the efficacy and safety of budesonide and formoterol fumarate metered dose inhaler relative to budesonide metered dose inhaler in adults and adolescents with inadequately controlled asthma.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, parallel group, multicenter study comparing Budesonide and Formoterol Fumarate Metered Dose Inhaler (BFF MDI) 160/9.6 μg twice daily (BID) to Budesonide MDI 160 μg (BD MDI), over 12 weeks. The study population will consist of adult and adolescent participants with asthma who remain inadequately controlled, as demonstrated by an Asthma Control Questionnaire (ACQ)-7 total score ≥1.5, despite treatment with low dose inhaled corticosteroid (ICS) or ICS/long-acting beta2-agonist (LABA). This study is to assess the benefits and safety of BFF MDI on lung function and asthma health-related quality of life.

This study will be conducted at approximately 90 sites worldwide and will randomize approximately 340 adult and adolescent participants.

ELIGIBILITY:
Inclusion Criteria

1. 12 to 80 years of age, male and female, BMI <40 kg/m2; females of childbearing potential should be using highly effective birth control.
2. Participants who have a documented history of physician-diagnosed asthma ≥ 6 months prior to Visit 1, according to GINA guidelines [GINA 2021]. Healthcare records for one year prior to Visit 1 must be provided for adolescent participants (12 to < 18 years of age) to ensure consistent evaluation and follow-up of treatment in those participants.
3. Participants who have been regularly using a stable daily ICS or an ICS/LABA regimen (including a stable ICS dose), with allowed ICS doses, for at least 8 weeks prior to Visit 1.
4. ACQ-7 total score ≥ 1.5 at Visits 1 and 4.
5. A pre-bronchodilator/pre-dose FEV1 < 90% predicted normal value at Visits 1, 2, and 3 and a pre-dose FEV1 of 50% to 90% at Visit 4 (pre-randomization).
6. Reversibility to albuterol, defined as a post-albuterol increase in FEV1 of ≥ 12% and ≥ 200 mL for participants ≥ 18 years of age OR a post-albuterol increase in FEV1 of ≥ 12% for participants 12 to < 18 years of age either in the 12 months prior to Visit 1 or at Visit 2 or Visit 3, if repeat testing is necessary.
7. A pre-bronchodilator/pre-dose FEV1 at Visits 2, 3, and 4 that has not changed 20% or more (increase or decrease) from the pre-bronchodilator/pre-dose FEV1 recorded at the previous visit.
8. Asthma stability during run-in based on Investigator discretion using the symptom worsening assessment defined in Section 8.1.2.8 as a guideline.
9. Willing and, in the opinion of the Investigator, able to adjust current asthma therapy, as required by the protocol.
10. Demonstrate acceptable MDI administration technique.
11. eDiary compliance ≥ 70% during screening, defined as completing the daily eDiary and answering "Yes" to taking 2 puffs of run-in BD MDI for any 10 mornings and 10 evenings in the last 14 days prior to randomization.

Exclusion criteria

1. Life-threatening asthma as defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s).
2. Any respiratory infection or asthma exacerbation treated with systemic corticosteroids and/or additional ICS treatment in the 8 weeks prior to Visit 1 and throughout the Screening Period.
3. Hospitalization for asthma within 8 weeks of Visit 1.
4. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, hematological, neurological, endocrine, gastrointestinal, or pulmonary (eg, active tuberculosis, bronchiectasis, pulmonary eosinophilic syndromes, and COPD). Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or that could affect the efficacy or safety analysis.
5. Known history of drug or alcohol abuse within 12 months of Visit 1.
6. Unresectable cancer that has not been in complete remission for at least 5 years prior to Visit 1. Note: Squamous cell and basal cell carcinomas of the skin are not exclusionary.
7. Participation in another clinical study with a study intervention administered in the last 30 days or 5 half-lives, whichever is longer. Any other study intervention that is not identified in this protocol is prohibited for use during study duration.
8. Previous or current randomization into studies within the AEROSPHERE program including KALOS, LOGOS, VATHOS, LITHOS, or any glycopyrronium studies (PT001).
9. Use of a nebulizer or a home nebulizer for receiving asthma medications. Note: Acute use of a nebulizer for an asthma exacerbation during hospitalization is allowed as long as there is no occurrence within 8 weeks of Visit 1.
10. Do not meet the stable dosing period prior to Visit 1 or unable to abstain from protocol-defined prohibited medications during Screening and Treatment Periods.
11. Receipt of COVID-19 vaccine (regardless of vaccine delivery platform, eg, vector, lipid nanoparticle) ≤7 days prior to Visit 1 (from last vaccination or booster dose).
12. Participants with known hypersensitivity to beta2-agonists, corticosteroids, or any component of the MDI.
13. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, vital signs, or ECG, which in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study.
14. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months prior to Visit 1 (including all forms of tobacco, e-cigarettes or other vaping devices, and marijuana).
15. Planned hospitalization during the study.
16. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
17. Study Investigators, sub-Investigators, coordinators, and their employees or immediate family members.
18. Judgment by the Investigator that the participant is unlikely to comply with study procedures, restrictions and requirements.
19. For women only - currently pregnant (confirmed with positive highly sensitive urine pregnancy test), breast-feeding, or planned pregnancy during the study or not using acceptable contraception measures, as judged by the Investigator.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (57):
  - Research Site, Chandler, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Encinitas, California
  - Research Site, Fresno, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Ventura, California
  - Research Site, Walnut Creek, California
  - Research Site, Cutler Bay, Florida
  - Research Site, DeBary, Florida
  - Research Site, DeLand, Florida
  - Research Site, Miami, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, South Bend, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Rolla, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Missoula, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, New Windsor, New York
  - Research Site, Schenectady, New York
  - Research Site, Fayetteville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hatboro, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Boerne, Texas
  - Research Site, El Paso, Texas
  - Research Site, Forney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Victoria, Texas
  - Research Site, Waco, Texas
  - Research Site, American Fork, Utah
  - Research Site, Bountiful, Utah
  - Research Site, Milwaukee, Wisconsin
- Canada (9):
  - Research Site, Kamloops, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Winchester, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Czechia (7):
  - Research Site, Jindřichův Hradec
  - Research Site, Louny
  - Research Site, Lovosice
  - Research Site, Miroslav
  - Research Site, Prague
  - Research Site, Teplice
  - Research Site, Varnsdorf
- Malaysia (9):
  - Research Site, Alor Star
  - Research Site, George Town
  - Research Site, Ipoh
  - Research Site, Kajang
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Terengganu
  - Research Site, Sarawak Miri
  - Research Site, Seremban
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Marilao
- South Africa (4):
  - Research Site, Durban
  - Research Site, Newton
  - Research Site, Pretoria
  - Research Site, Tygervalley
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Guri-si
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5982C00005&attachmentIdentifier=23a99e44-8528-44a0-9f6f-75419ae20279&fileName=LITHOS_Clinical_Study_Report_Synopsis_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult and adolescent participants who have asthma which remains inadequately controlled (ACQ-7 total score ≥ 1.5) despite treatment with low dose ICS or ICS/LABA were recruited at 106 sites across 7 countries. Participants were randomized in a 1:1 scheme to BFF MDI 160/9.6 μg or BD MDI 160 μg. Randomization was stratified by baseline asthma treatment and age. The treatment period was 12 weeks in duration with up to 7 in-clinic visits during screening and treatment.
Pre-assignment Details: All participants had to be taking a stable daily low dose ICS or ICS/LABA for at least 8 weeks prior to Visit 1. After meeting the screening eligibility criteria, participants discontinued their low dose ICS or ICS/LABA at Visit 1 and initiated run-in BD MDI 160 µg taking BID until the evening prior to Visit 4 (randomization).
  Of the 374 randomized participants, all populations exclude 17 participants from 4 sites due GCP violation and 4 participants due to not receiving therapy.
Groups:
- BFF MDI 160/9.6 μg: Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg BID (320/19.2μg/day)
- BD MDI 160 μg: Budesonide (BD) metered-dose inhaler (MDI), 160 μg BID (320 μg/day)
Period: Overall Study
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Started | 179 | 174
Completed | 176 | 165
Not Completed | 3 | 9
Not completed — Failure to meet randomization criteria | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Population: The Efficacy Set is defined as all participants who are randomized to study intervention and receive any amount of randomized study intervention. It excludes 7 participants who were randomized before or concurrently in another study.
Groups:
- Total: Total of all reporting groups
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg | Total
Number analyzed (Participants) | 177 | 169 | 346
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (16.6) | 48.0 (16.1) | 48.4 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 128 | 241
  Male | 64 | 41 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 15 | 19 | 34
  Asian | 27 | 33 | 60
  White | 123 | 110 | 233
  Other | 10 | 5 | 15
  Multiple | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Global: Canada | 19 | 13 | 32
  Global: Czech Republic | 40 | 42 | 82
  Global: Malaysia | 4 | 5 | 9
  Global: Philippines | 11 | 11 | 22
  Global: South Africa | 11 | 15 | 26
  Global: South Korea | 3 | 3 | 6
  Global: United States | 89 | 80 | 169
Prior asthma medication [Count of Participants; unit: Participants]
  ICS | 43 | 42 | 85
  ICS/LABA | 134 | 127 | 261
Baseline reversibility (%) [Mean (Standard Deviation); unit: Percentage] — Reversibility (%) is calculated as (Post-Albuterol FEV1 - Pre-Albuterol FEV1)/Pre-Albuterol FEV1 x100
  Percentage | 21.8 (14.5) | 21.0 (14.6) | 21.4 (14.6)
Baseline pre-bronchodilator FEV1 (L) [Mean (Standard Deviation); unit: Liter] — Baseline pre-bronchodilator FEV1 (L) is the mean of the pre-dose FEV1 at -60 and -30 minutes on Day 1, using the best effort at each timepoint.
  Liter | 2.097 (0.630) | 2.047 (0.607) | 2.073 (0.619)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve 0 to 3 Hours (AUC0-3) at Week 12
Description: Change from baseline in forced expiratory volume in 1 second (FEV1) area under the curve 0 to 3 hours (AUC0-3) at Week 12. FEV1 AUC0-3 is calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time to report the result in liters. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 12
Population: The Efficacy Set is defined as all participants who are randomized to study intervention and receive any amount of randomized study intervention. Participants are analyzed according to the treatment assigned at randomization, regardless of the actual treatment received. Only subjects with non-missing baseline covariates used in the analysis model are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 175 | 168
Liter | 0.309 (0.0235) | 0.109 (0.0241)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.200, 95% CI 2-sided [0.134 to 0.267], Standard Error of Mean 0.0337 — An increase in estimate favors study drug. The model includes treatment, visit, prior maintenance medication, treatment-by-visit interaction, baseline trough FEV1, and percent Albuterol reversibility

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 at Week 12
Description: Change from baseline in morning pre-dose trough FEV1 at Week 12. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 175 | 168
Liter | 0.143 (0.0221) | 0.060 (0.0226)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p = 0.0096, ANCOVA; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.020 to 0.144], Standard Error of Mean 0.0316 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Onset of Action on Day 1: Absolute Change in FEV1 at 5 Minutes on Day 1
Description: Onset of action on Day 1: Absolute change in FEV1 at 5 minutes on Day 1. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: On Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 168 | 157
Liter | 0.179 (0.0138) | 0.026 (0.0142)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.153, 95% CI 2-sided [0.114 to 0.192], Standard Error of Mean 0.0198 — An increase in estimate favors study drug. The model includes treatment, timepoint, prior maintenance medication, treatment-by-timepoints interaction, baseline tFEV1, and % Albuterol reversibility

4. Secondary Outcome: Change From Baseline in the Mean Number of Puffs of Rescue Medication Use (Puffs/Day) Over 12 Weeks
Description: Change from baseline in the mean number of puffs of rescue medication use (puffs/day) over 12 Weeks. Baseline is the average during the last 7 days before randomization. Over 12 weeks is the average from randomization up to week 12. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: Over 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs/Day
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 171 | 167
Puffs/Day | -0.589 (0.0708) | -0.309 (0.0721)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p = 0.0058, ANCOVA; Mean Difference (Final Values) = -0.280, 95% CI 2-sided [-0.478 to -0.082], Standard Error of Mean 0.1008 — A decrease in estimate favors study drug. The model includes treatment, 4-week interval, their interaction, prior maintenance medication, severe asthma exacerbation history, baseline daily rescue use, baseline tFEV1, and % Albuterol reversibility

5. Secondary Outcome: Percentage of Responders in ACQ-7 (≥ 0.5 Decrease Equals Response) at Week 12
Description: Percentage of responders in ACQ-7 at Week 12, where responders are defined as participants with a ≥0.5 decrease in total score from baseline. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 175 | 168
Percentage of participants | 74.3 | 61.9
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p = 0.0101, Regression, Logistic; Odds Ratio (OR) = 1.851, 95% CI 2-sided [1.158 to 2.958] — An odds ratio greater than 1 favors study drug. The model includes treatment, prior maintenance medication, baseline instrument score, baseline tFEV1, and % Albuterol reversibility

6. Secondary Outcome: Percentage of Responders in ACQ-5 (≥ 0.5 Decrease Equals Response) at Week 12
Description: Percentage of responders in ACQ-5 at Week 12, where responders are defined as participants with a ≥0.5 decrease in total score from baseline. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 175 | 168
Percentage of participants | 77.1 | 62.5
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 2.114, 95% CI 2-sided [1.302 to 3.432] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Percentage of Responders in the Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(s) +12) (≥ 0.5 Increase Equals Response) at Week 12
Description: Percentage of responders in the Asthma Quality of Life Questionnaire for 12 years and older (AQLQ(s)+12) at Week 12, where responders are defined as participants with a ≥0.5 increase in total score from baseline. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 172 | 162
Percentage of participants | 61.6 | 47.5
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p = 0.0084, Regression, Logistic; Odds Ratio (OR) = 1.873, 95% CI 2-sided [1.175 to 2.985] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Rate of Severe Asthma Exacerbation (Pooled LITHOS and VATHOS Data) During the Treatment Period (up to 24 Weeks)
Description: As requested by a Health Authority, data from LITHOS and VATHOS (NCT05202262), two studies originally designed to assess lung function, were pooled to analyze the annualized rate of severe asthma exacerbations. This analysis was prespecified, uses data up to 12 weeks for LITHOS and 24 weeks for VATHOS, and was incorporated into the multiple testing procedure. An exacerbation is considered severe if it results in at least one of the following: a course of systemic corticosteroids (SCS) for ≥3 consecutive days to treat symptoms of asthma worsening, an ER or urgent care visit due to asthma requiring treatment with SCS, an in-patient hospitalization due to asthma, or death related to asthma. Treatment policy is implemented to handle all intercurrent events except for initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is used.
Time Frame: 24 Weeks
Population: The Efficacy Set is defined as all participants in LITHOS and VATHOS (NCT05202262) who are randomized to study intervention and receive any amount of randomized study intervention. Participants are analyzed according to the treatment assigned at randomization, regardless of the actual treatment received. Only subjects with non-missing baseline covariates used in the analysis model are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Exacerbations/year
Groups:
- BFF MDI 160/9.6 μg or 320/9.6 μg: Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 160/9.6 μg BID (320/19.2μg/day) or Budesonide/ Formoterol Fumarate (BFF) metered-dose inhaler (MDI), 320/9.6 μg BID (640/19.2μg/day)
- BD MDI 160 μg or 320 μg: Budesonide (BD) metered-dose inhaler (MDI), 160 μg BID (320 μg/day) or Budesonide (BD) metered-dose inhaler (MDI), 320 μg BID (640 μg/day)
Arm/Group | BFF MDI 160/9.6 μg or 320/9.6 μg | BD MDI 160 μg or 320 μg
Number analyzed (Participants) | 425 | 335
Exacerbations/year | 0.35 (0.05) | 0.42 (0.07)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg or 320/9.6 μg vs BD MDI 160 μg or 320 μg; The comparison of interest is the formoterol effect; Test type: Superiority; p = 0.3610, Regression, Negative Binomial; Rate Ratio = 0.82, 95% CI 2-sided [0.54 to 1.25] — A rate ratio below 1 favors study drug. The model includes budesonide dose, formoterol dose, study, severe asthma exacerbation history, prior maintenance medications, baseline tFEV1, % Albuterol reversibility, and region

9. Secondary Outcome: Rate of Severe Asthma Exacerbation During the Treatment Period (up to 12 Weeks)
Description: Annualized rate of severe asthma exacerbation during the treatment period (up to 12 Weeks). An asthma exacerbation will be considered severe if it results in at least one of the following: a course of systemic corticosteroids for at least 3 consecutive days to treat symptoms of asthma worsening, an ER or urgent care visit due to asthma that required treatment with systemic corticosteroids, an in-patient hospitalization due to asthma, or death related to asthma. Treatment policy is implemented to handle all intercurrent events with the exception of initiation of new asthma therapy or administration of prohibited medications thought to impact efficacy in conjunction with premature discontinuation of randomised study intervention, for which the composite strategy is implemented.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Exacerbations/year
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
Number analyzed (Participants) | 177 | 169
Exacerbations/year | 0.25 (0.08) | 0.52 (0.12)
Statistical Analysis 1: Comparison: BFF MDI 160/9.6 μg vs BD MDI 160 μg; Test type: Superiority; p = 0.0419, Regression, Negative Binomial; Rate Ratio = 0.48, 95% CI 2-sided [0.23 to 0.97] — A rate ratio lower than 1 favors study drug. The model includes treatment, severe asthma exacerbation history, prior maintenance medications, baseline tFEV1, % Albuterol reversibility, and region

ADVERSE EVENTS:
Time Frame: From the date of first dose of IP up to and including 1 day following the date of last IP dose, up to 12 weeks.
Description: Adverse events were reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative). The Investigator and any designees were responsible for detecting, documenting, and recording events that meet the definition of an AE.
  The Safety Set is defined as the Efficacy Set, but it also includes the 7 participants who were randomized multiple times at sites or studies.
Arm/Group | BFF MDI 160/9.6 μg | BD MDI 160 μg
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/179 | 0/174
Other Adverse Events (participants affected / at risk) | 9/179 | 9/174
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFF MDI 160/9.6 μg (N=179) | BD MDI 160 μg (N=174)
Nasopharyngitis (Infections and infestations) | 3 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT05755906/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT05755906/SAP_001.pdf